CLINICAL TRIAL: NCT07035392
Title: A Single-arm, Prospective, Multicenter Clinical Study of Adebrelimab in Combination With Chemotherapy Neoadjuvant Therapy to Resect Non-small Cell Lung Cancer
Brief Title: Adebrelimab + Chemotherapy as Neoadjuvant Therapy for Resectable NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhangzhou Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024KYZ432
Record Dates: First submitted 2025-05-22; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Adebrelimab (SHR-1316); NSCLC; Chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab in combination chemotherapy (Experimental)
  Interventions: Drug: Adebrelimab; Drug: chemotherapy

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab 1200mg，ivgtt，D1，Q3W
Drug: chemotherapy — Queue A (lung squamous cell carcinoma patients):
  Albumin paclitaxel 260mg/m2, ivgtt，D1 , Q3W Carboplatin AUC=5, D1，Q3W
  Queue B (lung adenocarcinoma patients):
  Pemetrexed 500 mg/m2, ivgtt，D1，Q3W Carboplatin AUC=5, D1，Q3W

SUMMARY:
This study is a single arm, prospective, multicenter clinical trial, and eligible patients will receive the following treatment regimen: Adebrelimab combined with chemotherapy.The study includes a screening period (from the signing of informed consent by the subjects to no more than 28 days before the first medication, imaging examinations are allowed to be performed within 28 days before the first medication, and tumor tissue biopsy is allowed to be archived within 6 months before the first medication), a treatment period (including neoadjuvant and surgical treatment), and a follow-up period (including safety follow-up and survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 70 years old, male or female not limited;
2. ECOG PS score 0-1 points;
3. Patients who have not received systematic treatment in the past and agree to undergo radical surgery; Patients without surgical contraindications judged by thoracic surgeons;
4. Stage II, IIIA, or selective IIIB (T3N2M0 only) squamous or non squamous cell non-small cell lung cancer confirmed by histopathology or cytology and judged by researchers to be capable of undergoing R0 surgical resection for the purpose of cure. Disease staging should be based on the American Joint Committee on Cancer (AJCC)/International Union Against Cancer (UICC) NSCLC staging system, 8th edition;
5. There is sufficient tumor tissue to detect PD-L1 expression level and PD-L1 ≥ 1%;
6. At least one measurable lesion (according to RECIST 1.1 criteria);
7. The expected survival period is at least 12 weeks;
8. Other major organs (liver, kidney, blood system, etc.) are functioning well:

   * Hemoglobin ≥ 90g/L (no blood transfusion, no use of hematopoietic factors, and no medication correction within 2 weeks before the first medication);
   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
   * Platelet count ≥ 100 × 109/L; Total bilirubin ≤ 1.5 times the upper limit of normal value;
   * alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase ≤ 2.5 times the upper limit of normal values;
   * Serum creatinine ≤ 1.5 times the upper limit of normal value; And the endogenous creatinine clearance rate is ≥ 60ml/min; For patients who have not received anticoagulant therapy, the international normalized ratio (INR) of prothrombin time is ≤ 1.5, and the activated partial thromboplastin time (APTT) is ≤ 1.5 times the upper limit of normal.
9. Expected to be completely resected;
10. Good lung function can tolerate surgical treatment;
11. Female participants with fertility must undergo a pregnancy test (serum or urine) within 72 hours before starting the study medication, and the result must be negative. They must also be willing to use a medically recognized and effective contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study period and within 90 days after the last administration of the study medication; For male participants whose partners are women of childbearing age, they must agree to use effective methods of contraception or have undergone surgical sterilization during the study period and within 90 days after the last study administration;
12. The subjects voluntarily joined this clinical study and signed an informed consent form.

Exclusion Criteria:

1. Previously received any anti-tumor treatment, including radiotherapy, chemotherapy, immunotherapy, and traditional Chinese medicine anti-tumor treatment (excluding treatment for malignant tumors that have been cured and have no recurrence or metastasis for ≥ 5 years);
2. Non squamous cell carcinoma histological types of NSCLC with EGFR mutation positive or ALK positive subjects. Non squamous cell carcinoma subjects must undergo EGFR gene testing and ALK gene and/or immunohistochemical testing;
3. Patients with distant metastases (including M1a, M1b, M1c);
4. Suffering from any active autoimmune disease or history of autoimmune disease (such as uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which can be included after hormone replacement therapy), tuberculosis); Skin diseases that have completely relieved childhood asthma and do not require any intervention or systemic treatment in adulthood (such as vitiligo, psoriasis, or hair loss) can be included, but patients who require medical intervention with bronchodilators cannot be included;
5. Exclude evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, imaging confirmed active pneumonia, and severe impairment of lung function;
6. Subjects who have received systemic therapy with corticosteroids (>10 mg/day of prednisone or other equivalent hormones) or other immunosuppressive agents within 2 weeks prior to their first administration. In the absence of active autoimmune diseases, inhalation or topical use of corticosteroids is allowed, as well as adrenal hormone replacement therapy with a dose of ≤ 10 mg/day effective dose of prednisone;
7. Imaging (CT or MRI) shows tumor invasion into large blood vessels or blurred boundaries with blood vessels; Or imaging (CT or MRI) shows the presence of any pulmonary cavities or necrotic lesions, as determined by the researcher;
8. Individuals who have experienced arterial/venous thrombotic events within the first 6 months of enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
9. Within the first 3 months of enrollment, there have been significant clinically significant bleeding symptoms or clear bleeding tendencies, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, etc., or they are currently receiving thrombolytic or anticoagulant therapy;
10. Prior to enrollment, there was a daily hemoptysis volume of 100mL or more or a high risk of hemoptysis determined by the researcher;
11. Individuals with hypertension who cannot achieve good control with antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg); Grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥ 450ms for males and ≥ 470ms for females); According to NYHA standards, patients with grade III-IV cardiac dysfunction or those with left ventricular ejection fraction (LVEF)<50% as indicated by cardiac ultrasound examination;
12. Individuals who have undergone other major surgeries or severe injuries within the two months prior to the start of this experiment;
13. Urine routine examination indicates urinary protein ≥ (++), or 24-hour urine protein level ≥ 1g, or severe liver and kidney dysfunction;
14. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
15. Allergic to the experimental drug;
16. Merge with HIV infection or active viral hepatitis;
17. Pregnant or lactating women; Subjects with fertility who are unwilling or unable to take effective contraceptive measures;
18. Individuals with neurological disorders or mental illnesses who are unable to cooperate;
19. Cervical carcinoma in situ, basal cell or squamous cell carcinoma that can be adequately treated, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery are excluded from concurrent malignant tumors occurring ≤ 5 years before enrollment;
20. Researchers believe that there are other situations that are not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Main pathological relief (MPR) | Four weeks after surgery
  Main pathological relief (MPR) is defined as less than or equal to 10% of active tumor tissue in the surgical specimen during tumor resection.

SECONDARY OUTCOMES:
pathologic complete response（pCR） | Four weeks after surgery
Surgical R0 resection rate | Four weeks after surgery
objective response rate(ORR) | Up to 3 months per two cycles (21 days per cycle)
The incidence and severity of adverse events (including serious adverse reactions) | Up to 24 weeks

IPD SHARING:
Plan to Share IPD: No